CLINICAL TRIAL: NCT06860308
Title: The Determination of the Effect of Norepinephrine Infusion on the Development of Pressure Injury Among Critically Ill Patients
Brief Title: The Effect of Norepinephrine on the Development of Pressure Injury
Status: Completed | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Ayda Kebapci, Associate Professor, Koç University
Other Study IDs: NR24022025
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Pressure Injury
Keywords: pressure injury; norepinephrine; vasopressor; intensive care; development
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case Group: Patients with norepinephrine infusion in the intensive care unit,
- Control group: Patients without norepinephrine in the intensive care unit

SUMMARY:
Norepinephrine mainly increases mean arterial pressure among intensive care patients. It may be an essential risk factor in developing pressure injuries. However, there are still conflicting findings in the literature.

This study aimed to examine the effect of norepinephrine infusion on the development of pressure injuries among patients in adult intensive care.

This retrospective and correlational study was conducted between March 2021- May 2022. The electronic patient data were obtained from 289 adult patients (Case group n=149; control group n=149) treated with and without norepinephrine in the intensive care unit, respectively. The demographic and clinical characteristics were evaluated using descriptive statistical methods (number, percentage, mean, standard deviation). A logistic regression model was established to estimate the dependent variable (development of pressure injury) with the independent variables.

ELIGIBILITY:
Inclusion Criteria:

The sample consisted of all patients

* over 18 years old
* who did not have pressure injuries upon admission to the intensive care unit. Patients who received norepinephrine and received norepinephrine infusion for at least 48 hours during their stay in ICU were included in the case group (n=149), and patients who did not receive an infusion were included in the control group (n=140).

Exclusion Criteria:

The sample excluded of all patients

* less than 18
* who have pressure injuries during admission
* who had norepinephrine infusion less than48 hours during their stay in the intensive care unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population included all adult critically ill patients hospitalized in the 16-bed Adult ICU at the university hospital in Istanbul, Turkey. The ICU was 3rd level ICU where medical and surgical patients received life support treatments and care at the highest level. The study was conducted between May 2020 and March 2021.
Sampling Method: Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
development of pressure injury after admission to intensive care unit until discharge | after admission of patients to the intensive care unit until discharge between from March 2021 to May 2022. .
  The development of pressure injuries after admission of patients to the intensive care unit until discharge between from March 2021 to May 2022. . This is a retrospective study, so there is no specific time. We specified time frame details below.

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data only can be shared during publication process with reviewer if necessary